CLINICAL TRIAL: NCT01520610
Title: Genetic Polymorphisms in Catecholamine Pathway Responsible for the Tako-TSUBO Cardiomyopathy Susceptibly (TAKO-GENE)
Brief Title: TAKO-TSUBO Cardiomyopathy and Genetic
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fédération Française de Cardiologie (Other)
Responsible Party: Sponsor
Other Study IDs: AOR 10018
Record Dates: First submitted 2011-12-23; First posted 2012-01-30 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-02

CONDITIONS: Tako-TSUBO Cardiomyopathy; Acute Coronary Syndrome
Keywords: Tako-TSUBO Cardiomyopathy; Stress Cardiomyopathy; Myocardiopathies; Acute Coronary Syndrome; Gene
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Acute Coronary Syndrome; Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 20 ml of blood sample will be collected from all patients enrolled in order to DNA analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- CTT: Patients with cardiopathy of tako TSUBO.
- SCA: Patients with acute coronary syndrome but without Tako-TSUBO cardiomyopathy.
- Surgical stress: patients with stressful event (emergency postoperative patients) but without Tako-TSUBO cardiomyopathy.

SUMMARY:
This is a case-control association study with multicentric prospective recruitment.

Tako-TSUBO cardiomyopathy is a new clinical entity mimicking an acute coronary syndrome. It is characterized by reversible left ventricular dysfunction that is frequently precipitated by a stressful event and most of patients are postmenopausal women.

Several hypotheses concerning pathogenesis of Tako-TSUBO cardiomyopathy have been proposed, but at present, exaggerated sympathetic stimulation is the main hypothesis. However, the investigators don't know why some patients with stressful event may present Tako-TSUBO cardiomyopathy whereas most of them don't.

The investigators hypothesize that polymorphisms in the genes involved in the adrenergic pathway resulting in greater catecholamine sensitivity would be associated with an increased risk of Tako-TSUBO cardiomyopathy.

DETAILED DESCRIPTION:
We hypothesize that polymorphisms in the genes involved in the adrenergic pathway resulting in greater catecholamine sensitivity would be associated with an increased risk of Tako-TSUBO cardiomyopathy.

Aim of this study:

Primary endpoint: Cognitive study aiming at identifying genetic polymorphisms in adrenergic pathway responsible for the Tako-TSUBO cardiomyopathy susceptibly.

Secondary endpoint: Study of clinical, ECG, angiographic, echocardiographic characteristics and outcome of patients presenting with Tako-TSUBO cardiomyopathy.

Methods:

Case-control association study with multicentric prospective recruitment. The study population will be consisted of 800 Caucasians subjects: 200 patients with Tako-TSUBO cardiomyopathy and an age- and sex-matched control group (n = 600) of 400 patients with acute coronary syndrome and 200 patients with stressful event (emergency postoperative patients) but without Tako-TSUBO cardiomyopathy. Sixteen candidates genes from the catecholamine pathway will be studied.

The diagnosis of Tako-TSUBO cardiomyopathy will be defined as (1) an acute chest pain during a stressful incident associated with ST-segment abnormalities and/or increased serum troponin level, (2) transient left ventricular systolic dysfunction, and (3) no coronary lesions related to the left ventricular dysfunction.

Diagnosis of acute coronary syndrome will be performed according to the definition of the American Heart Association/American College of Cardiology and European Society of Cardiology.

We will genotype all the known functional SNPs (Single Nucleotide Polymorphisms) and the Tag SNPs representative of at least 80% of the total genetic diversity (available at HapMap web site). SNPs will be studied alone or combined in haplotype.

ELIGIBILITY:
"Tako-TSUBO" group:

Inclusion criteria :

* Patients presenting with Tako-TSUBO cardiomyopathy defined as: 1) an acute chest pain during a stressful incident associated with ST-segment abnormalities and/or increased serum troponin level, 2) transient left ventricular systolic dysfunction, and 3) no coronary lesions related to the left ventricular dysfunction
* Age > 18
* Written consent
* Caucasian origin
* Affiliation to health care system

Exclusion criteria :

* Patients presenting with pheochromocytoma
* Patients presenting with myocarditis
* Patients presenting with subarachnoid hemorrhage

"Acute coronary syndrome" group (age- and sex-matched control group):

Inclusion criteria :

* Patients presenting with an acute coronary syndrome (according to the definitions of guidelines)
* Age > 18
* written consent
* Caucasian origin
* Affiliation to health care system

Exclusion criteria :

* Patients presenting with a suspicion of Tako-TSUBO cardiomyopathy
* Patients presenting with a history of Tako-TSUBO cardiomyopathy

"Surgical stress" group (age- and sex-matched control group):

Inclusion criteria :

* Patients hospitalized for an urgent surgery
* Age > 18
* Written consent
* Caucasian origin
* Affiliation to health care system

Exclusion criteria :

* Patients presenting with increase of troponin after surgery
* Patients presenting with ECG abnormalities after surgery
* Patients presenting with a suspicion of Tako-TSUBO cardiomyopathy
* Patients presenting with a history of Tako-TSUBO cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be consisted of 800 Caucasians subjects: 200 patients with Tako-Tsubo cardiomyopathy and an age- and sex-matched control group (n = 600) of 400 patients with acute coronary syndrome and 200 patients with stressful event (emergency postoperative patients) but without Tako-Tsubo cardiomyopathy.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
DNA analysis | 48 months
  To identify genetic polymorphisms in adrenergic pathway responsible for the Tako-TSUBO cardiomyopathy susceptibly

SECONDARY OUTCOMES:
Diagnosis and prognosis of Tako-TSUBO cardiomyopathy | 48 months
  To assess diagnostic criteria of Tako-TSUBO cardiomyopathy To assess the prognosis of Tako-TSUBO cardiomyopathy

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Mansencal, MD, PHD, Principal Investigator — Hôpitaux de Paris (AP-HP), Hôpital Ambroise Paré. Université de Versailles-Saint Quentin en Yvelines
Locations (1):
- Name: Assistance Publique - Hôpitaux de Paris (AP-HP), Hôpital Ambroise Paré. Université de Versailles-Saint Quentin en Yvelines, Boulogne-Billancourt, Hautes Des Seine, France